CLINICAL TRIAL: NCT05429112
Title: A Randomized Comparison Between the Flexible Tip Bougie Vs Tube with Stylet for First-attempt Intubation Success with a Videolaryngoscopy in ICU Patients
Brief Title: Flexible Tip Bougie Vs Tube with Stylet for Intubation with a Videolaryngoscopy in ICU (VIDEOL-FLEXTIP)
Acronym: VIFLEXTIPICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Professor, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VIDEOLAR-FLEXTIP-ICU
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Intubation; Difficult or Failed
Keywords: intubation; difficult airway; videolaryngoscope; Intensive Care Unit; bougie

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endotracheal Tube with Stylet (Active Comparator): Patients randomised to Endotracheal Tube with Stylet will be intubated with a Videolaryngoscopy and with a endotracheal tube + stylet.
  Interventions: Device: Endotracheal Tube with Stylet
- Flexible Tip Bougie (Active Comparator): Patients randomised to Flexible Tip Bougie will be intubated with a Videolaryngoscopy and with a Flexible Tip Bougie.
  Interventions: Device: Flexible Tip Bougie

INTERVENTIONS:
Device: Flexible Tip Bougie — Patients randomised to Flexible Tip Bougie will be intubated with a Videolaryngoscopy and with a Flexible Tip Bougie.
  Arms: Flexible Tip Bougie
Device: Endotracheal Tube with Stylet — Patients randomised to Endotracheal Tube with Stylet will be intubated with a Videolaryngoscopy and with a endotracheal tube + stylet.
  Arms: Endotracheal Tube with Stylet

SUMMARY:
Tracheal intubation in the intensive care unit (ICU) is associated with high incidence of difficult intubation and complications . Videolaryngoscopes (VLs) devices have been proposed to improve airway management, and the use of VLs are recommended as first-line or after a first-attempt failure using direct laryngoscopy in ICU airway management algorithms. Although two meta-analysis showed that videolaryngoscopy improves visualization of the glottis and the first-attempt success, other two meta-analysis reported that videolaryngoscopy didn´t improve first-attempt success rate. The reason may be that although VLs improve glottic visualization, on many occasions it may not be accompanied by intubation at the first attempt, because the endotracheal tube has to pass a sharp angle to enter the trachea. To avoid this limitation, a new flexible tip bougie is designed to flexibly navigate the distal tip and help facilitate precise insertion of the endotracheal tube in the trachea .

DETAILED DESCRIPTION:
Although VLs improve glottic visualization, on many occasions it may not be accompanied by intubation at the first attempt, because the endotracheal tube has to pass a sharp angle to enter the trachea. To avoid this limitation, a new flexible tip bougie is designed to flexibly navigate the distal tip and help facilitate precise insertion of the endotracheal tube in the trachea. The flexible tip bougie has an integrated slider along the surface which moves the tip anterior and posterior while the pre-curved distal portion of shaft allows the angulation to provide anterior flexion. This new flexible tip bougie could be used as a rescue when first intubation failure using the videolaryngoscopy, or as a first option to improve the percentage of patients intubated at the first attempt.

The purpose of this prospective randomized study is to compare successful intubation on the first attempt wuth the new flexible tip bougie versus endotracheal tube with stylet during intubation with videolaryngoscopy of critically ill adults in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the intensive care unit (ICU) and require mechanical ventilation through a tracheal tube.
* Adult (age ≥ 18 years)
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Refusal of study participation or to pursue the study by the patient
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Difference in the first attempt success rate (percentage) | during intubation
  To compare the difference in the first attempt success rate (percentage) of different techniques for tracheal intubation.

SECONDARY OUTCOMES:
Difference in the overall success rate (percentage) | during intubation
  To compare the difference overall success rate (percentage) of different techniques for tracheal intubation.
Difference in the incidence of complications related to intubation | Participants will be followed from the beginning of the intervention to 30 minutes after the intervention
  To compare the difference in complications (percentage) of different techniques for tracheal intubation:
  Hypoxemia (SpO2) < 90 %, Hypoxemia severe (SpO2) < 80 %, Hypotension defined as systolic blood pressure less than 80 mm Hg, Severe hypotension defined as systolic blood pressure less than 65 mm Hg, Cardiac arrest, death during intubation, Moderate or difficult intubation, oesophageal intubation, pulmonary aspiration, dental injuries.
Difficulty of intubation | during intubation
  Operator-assessed subjective difficulty of intubation by means of a special analogue numerical scale from 0 to 10, where 0=no subjective difficulty and 10=maximal subjective difficulty
Modified Cormack-Lehane grade of glottic view | during intubation
  Modified Cormack-Lehane grade of glottic view:
  I: full view of the glottis IIa: partial view of the glottis IIb: arytenoid or posterior part of the vocal cords just visible III: only epiglottis visible IV: neither glottis nor epiglottis visible
Additional airway equipment | during intubation
  Need for additional airway equipment
Number of intubation attempts | during intubation
  Number of intubation attempts

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada Muñiz, Ph.D., Principal Investigator — University Clinical Hospital of Santiago de Compostela
Locations (1):
- University Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data types: Deidentified participant data How to access data: Requests must be sent to manutabo@yahoo.es When available: With publication Additional Information Who can access the data: Researchers whose proposed use of the data has been approved T ypes of analyses: For scientific purpose Mechanisms of data availability: With investigator support
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When available: With publication
Access Criteria: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose

REFERENCES:
- [Background] Ruetzler K, Smereka J, Abelairas-Gomez C, Frass M, Dabrowski M, Bialka S, Misiolek H, Plusa T, Robak O, Aniolek O, Ladny JR, Gorczyca D, Ahuja S, Szarpak L. Comparison of the new flexible tip bougie catheter and standard bougie stylet for tracheal intubation by anesthesiologists in different difficult airway scenarios: a randomized crossover trial. BMC Anesthesiol. 2020 Apr 20;20(1):90. doi: 10.1186/s12871-020-01009-7. PMID 32312225
- [Background] Driver BE, Prekker ME, Klein LR, Reardon RF, Miner JR, Fagerstrom ET, Cleghorn MR, McGill JW, Cole JB. Effect of Use of a Bougie vs Endotracheal Tube and Stylet on First-Attempt Intubation Success Among Patients With Difficult Airways Undergoing Emergency Intubation: A Randomized Clinical Trial. JAMA. 2018 Jun 5;319(21):2179-2189. doi: 10.1001/jama.2018.6496. PMID 29800096
- [Background] Driver BE, Semler MW, Self WH, Ginde AA, Trent SA, Gandotra S, Smith LM, Page DB, Vonderhaar DJ, West JR, Joffe AM, Mitchell SH, Doerschug KC, Hughes CG, High K, Landsperger JS, Jackson KE, Howell MP, Robison SW, Gaillard JP, Whitson MR, Barnes CM, Latimer AJ, Koppurapu VS, Alvis BD, Russell DW, Gibbs KW, Wang L, Lindsell CJ, Janz DR, Rice TW, Prekker ME, Casey JD; BOUGIE Investigators and the Pragmatic Critical Care Research Group. Effect of Use of a Bougie vs Endotracheal Tube With Stylet on Successful Intubation on the First Attempt Among Critically Ill Patients Undergoing Tracheal Intubation: A Randomized Clinical Trial. JAMA. 2021 Dec 28;326(24):2488-2497. doi: 10.1001/jama.2021.22002. PMID 34879143
- [Background] Jaber S, Rolle A, Godet T, Terzi N, Riu B, Asfar P, Bourenne J, Ramin S, Lemiale V, Quenot JP, Guitton C, Prudhomme E, Quemeneur C, Blondonnet R, Biais M, Muller L, Ouattara A, Ferrandiere M, Saint-Leger P, Rimmele T, Pottecher J, Chanques G, Belafia F, Chauveton C, Huguet H, Asehnoune K, Futier E, Azoulay E, Molinari N, De Jong A; STYLETO trial group. Effect of the use of an endotracheal tube and stylet versus an endotracheal tube alone on first-attempt intubation success: a multicentre, randomised clinical trial in 999 patients. Intensive Care Med. 2021 Jun;47(6):653-664. doi: 10.1007/s00134-021-06417-y. Epub 2021 May 25. PMID 34032882